CLINICAL TRIAL: NCT01399372
Title: Phase II Randomized Study of Rituximab, Methotrexate, Procarbazine, Vincristine, and Cytarabine With and Without Low-Dose Whole-Brain Radiotherapy for Primary Central Nervous System Lymphoma
Brief Title: Rituximab, Methotrexate, Vincristine Sulfate, Procarbazine Hydrochloride, and Cytarabine With or Without Radiation Therapy in Treating Patients With Primary Central Nervous System Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 1114; CDR0000703682; NCI-2011-02678 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-07-20; First posted 2011-07-21 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-05

CONDITIONS: Chemotherapeutic Agent Toxicity; Cognitive/Functional Effects; Lymphoma; Neurotoxicity; Radiation Toxicity
Keywords: neurotoxicity; chemotherapeutic agent toxicity; radiation toxicity; cognitive/functional effects; primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Neurotoxicity Syndromes; Radiation Injuries | interventions — Rituximab; Cytarabine; Methotrexate; Procarbazine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy (Active Comparator): Rituximab, methotrexate, procarbazine for four 28-day cycles with vincristine for the first two cycles, followed 3-5 weeks later by two 28-day cycles of cytarabine.
  Interventions: Biological: Rituximab; Drug: Cytarabine; Drug: Methotrexate; Drug: Procarbazine; Drug: Vincristine
- Chemotherapy + Low-Dose WBRT (Experimental): Rituximab, methotrexate, procarbazine for four 28-day cycles with vincristine for the first two cycles, followed 2-5 weeks later by 3 weeks of low-dose whole-brain radiotherapy (WBRT), followed 3-5 weeks later by two 28-day cycles of cytarabine.
  Interventions: Biological: Rituximab; Drug: Cytarabine; Drug: Methotrexate; Drug: Procarbazine; Drug: Vincristine; Radiation: low-dose whole-brain radiation therapy

INTERVENTIONS:
Biological: Rituximab — One 28-day cycle = 500 mg/m^2 intravenously on day 1 and day 5.
Drug: Cytarabine — One 28-day cycle = 3 g/m^2 intravenously on day 1 and day 2.
Drug: Methotrexate — One 28-day cycle = 3.5 g/m^2 intravenously (standard hydration/leucovorin support) on day 2.
  Other Names: MTX
Drug: Procarbazine — One 28-day cycle = 100 mg/m^2 orally on days 2-8.
Drug: Vincristine — One 28-day cycle = 1.4 mg/m^2 intravenously, dose capped at 2.4mg, on day 2 and day 16.
Radiation: low-dose whole-brain radiation therapy — Total dose of 2340 cGy administered as 13 daily fractions of 180 cGy over 3 weeks. Participants with progressive disease on magnetic resonance imaging (MRI) do not receive WBRT.
  Other Names: WBRT
  Arms: Chemotherapy + Low-Dose WBRT

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and help kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as methotrexate, vincristine sulfate, procarbazine hydrochloride, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x rays to kill cancer cells. It is not yet know whether rituximab and combination chemotherapy are more effective when given with or without radiation therapy in treating patients with primary central nervous system lymphoma.

PURPOSE: This randomized phase II trial studies how well giving rituximab and combination chemotherapy with or without radiation therapy works in treating patients with primary central nervous system lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine median progression-free survival (PFS) in both arms on an intent-to-treat basis.

Secondary

* To determine overall survival (OS) defined as the interval from randomization to death due to any cause.
* To determine treatment-related neurotoxicity rates and disease-related cognitive deterioration in each arm, through the following methods: prospective formal neuropsychological evaluation, utilizing competing-risk methodology to account for death as a competing risk to neurotoxicity or cognitive deterioration from relapsed tumor burden/salvage treatment and incidence of clinically defined neurotoxicity as per investigator's assessment.
* To determine if there exists differences between the two treatment arms in terms of health-related quality-of-life and symptoms over time.
* To determine response (partial response (PR) and complete response (CR)) rate after methotrexate-based chemotherapy and after consolidation whole-brain radiotherapy (WBRT).
* To determine chemotherapy-related toxicity, measured by Common Toxicity Criteria for Adverse Effects (CTCAE), v.4.0.

OUTLINE: This is a multicenter study. Patients are stratified according to Memorial Sloan-Kettering Cancer Center recursive-partitioning analysis (RPA) classification for primary central nervous system lymphoma on age and Karnofsky performance status (KPS) (Class 1: age ≤ 50 years vs Class 2: age > 50 years and KPS ≥ 70% vs Class 3: age > 50 years and KPS < 70%). Patients are randomized to 1 of 2 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. B-cell non-Hodgkin's lymphoma(NHL) involving the brain, as demonstrated by contrast-enhanced Magnetic resonance imaging (MRI) and histologic confirmation by one of the following within 6 weeks prior to registration:

   * A positive cerebral spinal fluid (CSF) cytology for lymphoma or a monoclonal lymphocyte population as defined by cell surface markers
   * A biopsy of the vitreous or uvea demonstrating non-Hodgkin's lymphoma
   * Brain biopsy

   Note: Patients in whom the type of lymphoma could not be determined or is unknown (eg, not enough tissue for further analysis) are assumed to have a B cell lymphoma and are eligible.
2. The patient must agree to submit tissue (i.e., the original H/E stained slides and immunohistochemistry studies) for central pathology review post-registration.
3. No evidence of systemic non-Hodgkin lymphoma as demonstrated by a computed tomography (CT) scan of the chest, abdomen and pelvis within 6 weeks prior to registration (Note: Bone marrow biopsy is not required for registration but must be obtained prior to start of treatment.)
4. Age ≥ 18
5. History and physical examination within 6 weeks of registration
6. Karnofsky performance status (KPS) equal to 50 or higher, with the following exception

   • Patients with KPS 30 to 50 are eligible if the reason for the poor performance status is neurologic deficit from primary central nervous system (CNS) lymphoma. (Patients with KPS 30 to 50 due to reasons other than primary CNS lymphoma are ineligible. Patients with KPS under 30 for any reason are ineligible)
7. Patient must have documentation of negative HIV-1 testing within 6 weeks prior to study registration (Separate counseling and consent as per institutional guidelines)
8. Complete blood count (CBC)/differential obtained within 2 weeks prior to study registration, with adequate bone marrow function defined as follows:

   * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3;
   * Platelets ≥ 100,000 cells/mm3;
   * Hemoglobin (Hgb) ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.);
9. Adequate liver function within 2 weeks prior to study registration, defined as follows:

   * Bilirubin < 2.0 mg/dl
   * Aspartate aminotransferase (AST) <2.5 times upper limit of normal
10. Adequate renal function within 2 weeks prior to study registration, defined as follows

    * Serum creatinine < 1.5 mg/dl
    * Calculated creatinine clearance (CrCl) > 50cc/min/1.73m2, using the Cockcroft-Gault equation, as follows:

    Male: CrCl (ml/min) = (140-age) X (Actual weight in kg) / 72 x serum Creatinine (mg/dl).

    Female: CrCl (ml/min) = (140-age) X (Actual weight in kg) X 0.85 / 72 x serum Creatinine (mg/dl).

    Note: A measured CrCl from a 24 hour urine collection may also be used.
11. Women of childbearing potential and male participants must agree to practice adequate contraception during therapy
12. Patient must provide study-specific informed consent prior to study registration
13. Patient must be able to swallow pills.

Exclusion Criteria:

1. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
2. Prior treatment with chemotherapy or radiotherapy for lymphoma or chronic lymphocytic leukemia; note that prior chemotherapy for a different cancer is allowable; see section 1
3. Prior cranial irradiation
4. Severe, active co-morbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
   * Transmural myocardial infarction within the last 6 months;
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
   * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration
   * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
   * Known pre-existing immunodeficiency as seen in organ transplant recipient.
5. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
6. Prior allergic reaction to any of the study drugs involved in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-09; Primary Completion 2020-03-19 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Omuro, MD, Principal Investigator — Yale University
Locations (45):
- United States (44):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Oncology-Deer Valley Center, Phoenix, Arizona
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cadence Cancer Center in Warrenville, Warrenville, Illinois
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center Commack, Commack, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University Pointe, West Chester, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - American College of Radiology Imaging Network, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - M D Anderson Cancer Center CCOP Research Base, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemotherapy | Chemotherapy + Low-Dose WBRT
Started | 47 | 44
Eligible | 44 | 43
Eligible and Started Protocol Treatment | 43 | 43
Completed (Participants contributing data to results are considered to have completed the study) | 44 | 43
Not Completed | 3 | 1
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy | Chemotherapy + Low-Dose WBRT | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Customized [Median (Full Range); unit: years] | 59.5 [21 to 84] | 66 [40 to 78] | 63 [21 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 22 | 23 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 38 | 37 | 75
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 33 | 37 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Karnofsky Performance Status (KPS) [Count of Participants; unit: Participants] — 30 = Severely disabled, hospitalization is indicated, although death not imminent; 40 = Disabled, requires special care and assistance; 50 = Requires considerable assistance and frequent medical care; 60 = Requires occasional assistance, but is able to care for most personal needs; 70 = Cares for self, unable to carry on normal activity or to do active work; 80 = Normal activity with effort, some signs or symptoms of disease; 90 = Able to carry on normal activity, minor signs or symptoms of disease; 100 = Normal no complaints, no evidence of disease.
  Participants
    30-50 | 5 | 6 | 11
    60-80 | 23 | 22 | 45
    90-100 | 16 | 15 | 31
Neurologic Symptoms [Count of Participants; unit: Participants]
  None | 8 | 7 | 15
  Minor | 15 | 16 | 31
  Moderate | 18 | 14 | 32
  Severe | 3 | 6 | 9
Memorial Sloan-Kettering Cancer Center (MSKCC) Recursive Partitioning analysis (RPA) Class [Count of Participants; unit: Participants] — Class 1: age <= 50; class 2: age >50 and KPS >=70; class 3: age > 50 and KPS <70
  Participants
    Class 1 | 7 | 6 | 13
    Class 2 | 26 | 25 | 51
    Class 3 | 11 | 12 | 23
Ocular Involvement [Count of Participants; unit: Participants] | 3 | 0 | 3
Cerebrospinal fluid (CSF) Involvement [Count of Participants; unit: Participants] | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression is defined as any of the following: more than 25% increase in the contrast-enhancing lesion seen on magnetic resonance imaging (MRI) compared with baseline or best response; new site of disease (central nervous system or systemic); recurrent or new ocular disease; recurrent or positive cerebrospinal fluid (CSF) cytology. Progression-free survival time is defined as time from randomization to the date of first progression, death, or last known follow-up (censored). Progression-free survival rates are estimated using the Kaplan-Meier method.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 7.3 years.
Population: Eligible participants
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Chemotherapy | Chemotherapy + Low-Dose WBRT
Number analyzed (Participants) | 44 | 43
years | 2.1 [1.0 to NA] — There were not enough events to estimate the upper confidence boundary. | NA [3.3 to NA] — The median has not yet been reached. Additionally there were not enough events to estimate the upper confidence boundary.
Statistical Analysis 1: Comparison: Chemotherapy vs Chemotherapy + Low-Dose WBRT; Sample size of 89 provided 80% power to detect a hazard ratio of 0.63 at a one-sided alpha level of 0.15; Test type: Superiority; p = 0.015, Log Rank — One-sided significance level = 0.15; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.27 to 0.95] — Reference arm = Chemotherapy

2. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 7.3 years.
Population: Eligible participants
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Chemotherapy | Chemotherapy + Low-Dose WBRT
Number analyzed (Participants) | 44 | 43
years | NA [2.6 to NA] — The median has not yet been reached. Additionally there were not enough events to estimate the upper confidence boundary. | NA [4.5 to NA] — The median has not yet been reached. Additionally there were not enough events to estimate the upper confidence boundary.
Statistical Analysis 1: Comparison: Chemotherapy vs Chemotherapy + Low-Dose WBRT; Test type: Superiority; p = 0.48, Log Rank — Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.38 to 1.58] — Reference arm = Chemotherapy

3. Secondary Outcome: Percentage of Participants Experiencing Partial Response or Complete Response
Description: Response was evaluated using the international criteria proposed by the International Primary Central Nervous System Lymphoma (PCNSL) Study Group criteria. Complete Response was defined as no contrast brain enhancement on magnetic resonance imaging (MRI), no corticosteroid use for at least 2 weeks, a normal eye exam, and negative CSF cytology. Partial response was defined as at least 50% decrease in enhancing tumor on MRI compared with baseline imaging, no or minor retinal pigment epithelium (RPE) abnormality, and negative CSF cytology.
Time Frame: After 4th cycle of chemotherapy, approximately 4 months after randomization.
Population: Eligible participants with Cycle 4 disease assessment data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy | Chemotherapy + Low-Dose WBRT
Number analyzed (Participants) | 30 | 31
percentage of participants | 83.3 [65.3 to 94.4] | 80.6 [62.5 to 92.5]

4. Secondary Outcome: Global Heath Status (GHS) Score of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: Global Health Status is calculated from two questions on the EORTC QLQ-C30. The question responses range from 1 "very poor" to 7 "excellent" such that a higher response indicates better quality of life (QOL). The mean of these responses is linearly transformed to a range of 0 (worst) to 100 (best). Data through five years after end of protocol treatment is included in the analysis, while summary data is provided only through three years due to very few participants after that timepoint.
Time Frame: EORTC QLQ-C30 was administered at baseline, after cycle 4 of treatment (4 months), then every six months after end of treatment (7 months) for five years.
Population: Eligible, consented to quality of life study component, and has GHS score for at least one timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chemotherapy | Chemotherapy + Low-Dose WBRT
Number analyzed (Participants) | 34 | 35
score on a scale
  Baseline: number analyzed (Participants) | 30 | 34
  Baseline | 62.78 (23.54) | 54.90 (26.91)
  End of cycle 4: number analyzed (Participants) | 25 | 28
  End of cycle 4 | 67.67 (23.97) | 64.58 (20.49)
  6 Months Post-Treatment: number analyzed (Participants) | 18 | 24
  6 Months Post-Treatment | 74.54 (20.70) | 75.35 (20.48)
  12 Months Post-Treatment: number analyzed (Participants) | 12 | 23
  12 Months Post-Treatment | 78.47 (22.88) | 78.99 (24.73)
  18 Months Post-Treatment: number analyzed (Participants) | 14 | 20
  18 Months Post-Treatment | 76.79 (20.46) | 76.67 (24.27)
  24 Months Post-Treatment: number analyzed (Participants) | 12 | 14
  24 Months Post-Treatment | 70.83 (25.00) | 83.33 (21.43)
  30 Months Post-Treatment: number analyzed (Participants) | 12 | 18
  30 Months Post-Treatment | 77.08 (24.13) | 79.63 (17.90)
  36 Months Post-Treatment: number analyzed (Participants) | 10 | 15
  36 Months Post-Treatment | 75.00 (27.78) | 85.00 (13.80)
  42 Months Post-Treatment: number analyzed (Participants) | 4 | 13
  42 Months Post-Treatment | 75.00 (21.52) | 77.56 (19.95)
  48 Months Post-Treatment: number analyzed (Participants) | 7 | 8
  48 Months Post-Treatment | 79.76 (21.97) | 84.38 (19.64)
  54 Months Post-Treatment: number analyzed (Participants) | 7 | 5
  54 Months Post-Treatment | 70.24 (16.67) | 91.67 (10.21)
  60 Months Post-Treatment: number analyzed (Participants) | 3 | 1
  60 Months Post-Treatment | 80.56 (17.35) | 83.33 (NA) — Standard deviation cannot be computed if there is only one observation, as in this case.
Statistical Analysis 1: Comparison: Chemotherapy vs Chemotherapy + Low-Dose WBRT; A mixed effects model of EORTC QLQ-C30 GHS was run with independent variables treatment arm, time, baseline Memorial Sloan-Kettering Cancer Center (MSKCC) recursive partitioning analysis (RPA) class, and baseline neurologic symptoms (none/minor vs. moderate/severe), including the interaction of treatment and time, representing difference in the longitudinal trajectory of the scores between the treatment arms. Prospectively, the interaction effect was of most interest and is reported here,; Test type: Superiority; p = 0.005, Mixed Models Analysis

5. Secondary Outcome: Percentage of Participants With Neurocognitive Failure
Description: Neurocognitive failure is defined as cognitive failure on two or more of the following tests: Hopkins Verbal Learning Test - Revised (HVLT-R) Free Recall, HVLT-R Delayed Recall, HVLT-R Delayed Recognition, Trail Making Test Part A, Trail Making Test Part B, and Controlled Oral Word Association. Cognitive failure for each test is defined as a change from baseline in raw score (post baseline score - baseline score) at or exceeding the minimally important difference reported in the literature [determined by the reliable change index (RCI) method] of -5, -3, -2,12, 26, and -12, respectively, indicating a worsening of neurocognitive function. Time to neurocognitive failure is defined as time from randomization to date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rates are estimated using the cumulative incidence method and the distributions of failure times are compared between the arms. Two-year estimates are provided here.
Time Frame: Neurocognitive function tests were administered at baseline, after cycle 4 of treatment (4 months), then every six months after end of treatment (7 months) for five years. Two-year rates are provided here.
Population: Eligible, consented to neurocognitive function study component and has at least two completed neurocognitive tests at baseline and at least one post baseline visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy | Chemotherapy + Low-Dose WBRT
Number analyzed (Participants) | 30 | 32
percentage of participants | 31.6 [14.3 to 50.5] | 17.9 [6.3 to 34.1]
Statistical Analysis 1: Comparison: Chemotherapy vs Chemotherapy + Low-Dose WBRT; Test type: Superiority; p = 0.18, Gray's test; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.21 to 1.31] — Reference arm = Chemotherapy arm

6. Secondary Outcome: Distribution of Participants by Highest Grade Adverse Event Related to Protocol Treatment
Description: Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data. Adverse events reported as definitely, probably, or possibly related to protocol treatment are considered to be related to treatment.
Time Frame: At the end of each chemotherapy 28-day cycle, then every 2 months for two years starting 4 weeks after treatment, then every 6 months for 3 years, then yearly. Maximum follow-up at time of analysis was 7.3 years.
Population: Eligible participants who started protocol treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy | Chemotherapy + Low-Dose WBRT
Number analyzed (Participants) | 43 | 43
Participants
  None | 2 | 3
  Grade 1 | 3 | 6
  Grade 2 | 4 | 5
  Grade 3 | 20 | 15
  Grade 4 | 14 | 13
  Grade 5 | 0 | 1

ADVERSE EVENTS:
Time Frame: At the end of each chemotherapy 28-day cycle, then every 2 months for two years starting 4 weeks after treatment, then every 6 months for 3 years. Maximum follow-up at time of analysis was 7.3 years.
Description: All-cause mortality was assessed in eligible participants. Adverse events were assessed in eligible participants who started protocol treatment.
Arm/Group | Chemotherapy | Chemotherapy + Low-Dose WBRT
All-Cause Mortality (participants affected / at risk) | 3/44 | 1/43
Serious Adverse Events (participants affected / at risk) | 22/43 | 21/43
Other Adverse Events (participants affected / at risk) | 42/43 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=43) | Chemotherapy + Low-Dose WBRT (N=43)
Anemia (Blood and lymphatic system disorders) | 6 | 5
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Heart failure (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Death NOS (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 1 | 2
Hypothermia (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 5 | 1
Sepsis (Infections and infestations) | 3 | 1
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 0 | 2
Investigations - Other (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 3 | 5
Platelet count decreased (Investigations) | 5 | 1
White blood cell decreased (Investigations) | 4 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0
Edema cerebral (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Nervous system disorders - Other (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypotension (Vascular disorders) | 3 | 0
Thromboembolic event (Vascular disorders) | 2 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=43) | Chemotherapy + Low-Dose WBRT (N=43)
Anemia (Blood and lymphatic system disorders) | 34 | 30
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 3 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3
Sinus tachycardia (Cardiac disorders) | 3 | 2
Hearing impaired (Ear and labyrinth disorders) | 1 | 4
Blurred vision (Eye disorders) | 7 | 5
Eye disorders - Other (Eye disorders) | 6 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 21 | 21
Diarrhea (Gastrointestinal disorders) | 8 | 9
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 | 3
Mucositis oral (Gastrointestinal disorders) | 7 | 4
Nausea (Gastrointestinal disorders) | 23 | 15
Vomiting (Gastrointestinal disorders) | 8 | 6
Chills (General disorders) | 4 | 0
Edema limbs (General disorders) | 12 | 5
Fatigue (General disorders) | 31 | 38
Fever (General disorders) | 7 | 5
Gait disturbance (General disorders) | 3 | 5
Infusion related reaction (General disorders) | 4 | 0
Pain (General disorders) | 10 | 7
Infections and infestations - Other (Infections and infestations) | 1 | 4
Mucosal infection (Infections and infestations) | 3 | 4
Skin infection (Infections and infestations) | 2 | 4
Upper respiratory infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 4 | 9
Bruising (Injury, poisoning and procedural complications) | 1 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 5
Activated partial thromboplastin time prolonged (Investigations) | 1 | 4
Alanine aminotransferase increased (Investigations) | 28 | 25
Alkaline phosphatase increased (Investigations) | 16 | 20
Aspartate aminotransferase increased (Investigations) | 25 | 22
Blood bilirubin increased (Investigations) | 6 | 6
Creatinine increased (Investigations) | 6 | 15
Investigations - Other (Investigations) | 6 | 6
Lymphocyte count decreased (Investigations) | 20 | 22
Neutrophil count decreased (Investigations) | 19 | 20
Platelet count decreased (Investigations) | 27 | 26
Weight gain (Investigations) | 4 | 5
Weight loss (Investigations) | 4 | 6
White blood cell decreased (Investigations) | 22 | 22
Anorexia (Metabolism and nutrition disorders) | 12 | 9
Hypercalcemia (Metabolism and nutrition disorders) | 6 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 19 | 15
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 7
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 3
Hypernatremia (Metabolism and nutrition disorders) | 7 | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 | 19
Hypocalcemia (Metabolism and nutrition disorders) | 14 | 19
Hypoglycemia (Metabolism and nutrition disorders) | 5 | 7
Hypokalemia (Metabolism and nutrition disorders) | 20 | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 2
Hyponatremia (Metabolism and nutrition disorders) | 11 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 4
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 7
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 3 | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 5 | 2
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 8
Ataxia (Nervous system disorders) | 4 | 2
Cognitive disturbance (Nervous system disorders) | 4 | 5
Dizziness (Nervous system disorders) | 8 | 4
Dysarthria (Nervous system disorders) | 2 | 3
Dysgeusia (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 16 | 19
Lethargy (Nervous system disorders) | 0 | 3
Memory impairment (Nervous system disorders) | 5 | 9
Paresthesia (Nervous system disorders) | 7 | 4
Peripheral motor neuropathy (Nervous system disorders) | 4 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 17 | 13
Seizure (Nervous system disorders) | 3 | 5
Agitation (Psychiatric disorders) | 5 | 2
Anxiety (Psychiatric disorders) | 11 | 11
Confusion (Psychiatric disorders) | 4 | 5
Depression (Psychiatric disorders) | 8 | 4
Insomnia (Psychiatric disorders) | 13 | 10
Acute kidney injury (Renal and urinary disorders) | 3 | 4
Hematuria (Renal and urinary disorders) | 3 | 1
Proteinuria (Renal and urinary disorders) | 2 | 4
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 3
Urinary frequency (Renal and urinary disorders) | 7 | 2
Urinary incontinence (Renal and urinary disorders) | 3 | 4
Urinary retention (Renal and urinary disorders) | 4 | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 5
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 3
Hypertension (Vascular disorders) | 7 | 4
Hypotension (Vascular disorders) | 3 | 1
Thromboembolic event (Vascular disorders) | 7 | 2

LIMITATIONS AND CAVEATS:
A planned interim efficacy analysis was performed after 42 events (death or progression). The final analysis was planned to occur after 67 events. The Data Monitoring Committee (DMC) recommended releasing the interim results for early reporting and these results are considered the final study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT01399372/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT01399372/ICF_001.pdf